CLINICAL TRIAL: NCT01023009
Title: Postoperative Evolution After Small Gauge Vitrectomy Without Eye Occlusion
Acronym: Vitrectomy
Status: Terminated | Type: Observational
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Other Study IDs: APEC0006
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Vitrectomy
Keywords: Occlusion; vitrectomy; small gauge vitrectomy; Postoperative occlusion
MeSH Terms: conditions — Bites and Stings | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eye occlusion
  Interventions: Procedure: vitrectomy

INTERVENTIONS:
Procedure: vitrectomy

SUMMARY:
After an uneventfully small gauge vitrectomy we don´t think is necessary to occlude the eye for 24 hours

ELIGIBILITY:
Inclusion Criteria:

* All patients with uneventful vitrectomy

Exclusion Criteria:

* Complicated vitrectomy or corneal lesion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients in inmediate postoperative vitreorretinal surgery without any complications
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Martinez-Castellanos, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, México, Mexico